CLINICAL TRIAL: NCT00327795
Title: Staged Approach to Coarctation and VSD Can Offer Optimal Outcomes
Brief Title: Surgical Outcomes in Pediatric Patients With Coarctation and VSD
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 06-010
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Diagnosis of Coarctation of the Aorta and VSD; Surgical Repair at CHOA; Between January 1, 2002 and December 31, 2005
Keywords: congenital heart disease; pediatric; surgical outcomes
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Recently, a paper was published that compared outcomes of patients requiring repair of aortic coarctation and ventricular septal defect. Some surgeons opt to repair both defects in one surgery while other surgeons do the repair in two separate operations. Recently at Children's Healthcare of Atlanta, we have adopted the practice of correcting both defects during the same operation but through two separate incisions (one on the chest and the other through the ribs on the side. This reduces the amount of time the patient is on the heart-lung bypass machine during surgery. This study is a review of patient charts to compare outcomes of patients who have had surgery to repair their coarctation and VSD during 2002 through 2005.

DETAILED DESCRIPTION:
This study is a retrospective chart review of patients who carry the diagnosis of aortic coarctation and VSD and have had their surgical repair at Children's Healthcare of Atlanta between the dates of January 1, 2002 and December 31, 2005. The data collected will be surgical data such as type of repair, and the time the patient required cross clamp, circulatory arrest and cardiopulmonary bypass while in the operating room for the repair(s). We would also like to gather post-operative information such as time the patient required ventilation, whether they required a re-operation during the same admission, along with intensive care hours and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of coarctation and VSD
* surgical repair at Children's Healthcare of Atlanta between January 1, 2002 and December 31, 2005.

Exclusion Criteria:

* does not have coarctation and VSD
* did not have surgery at Children's Healthcare of Atlanta between January 1, 2002 and December 31, 2005.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diagnosis of coarctation and VSD
Sampling Method: Non-Probability Sample
Enrollment: 32
Dates: Start 2006-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States